CLINICAL TRIAL: NCT02860663
Title: Effect of Different Vitamin D Vitamers on Vitamin D Status and Biomarkers for Bone Health and Cardiovascular Risk in Healthy Humans
Brief Title: Effect of Different Vitamin D Vitamers on Vitamin D Status
Acronym: VitD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KF 01 322182
Record Dates: First submitted 2016-07-19; First posted 2016-08-09 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Vitamin D Status
MeSH Terms: interventions — Cholecalciferol; Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin D3 (Active Comparator): 10 ug/d of vitamin D3 for 6 weeks
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D2 (Active Comparator): 10 ug/d of vitamin D2 for 6 weeks
  Interventions: Dietary Supplement: Vitamin D2
- 25OHD (Active Comparator): 10 ug/ of 25OHD for 6 weeks
  Interventions: Dietary Supplement: 25OHD

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 10 ug/d of vitamin D3 for 6 weeks
  Arms: Vitamin D3
Dietary Supplement: Vitamin D2 — 10 ug/d of vitamin D3 for 6 weeks
  Arms: Vitamin D2
Dietary Supplement: 25OHD — 10 ug/d of vitamin D3 for 6 weeks
  Arms: 25OHD

SUMMARY:
Background: Dietary intake of vitamin D includes vitamin D3 (VitD3), 25-hydroxyvitamin D3 (25OHD3) and vitamin D2 (VitD2). However, the bioactivity of the different species is currently not scientifically established.

Objective: The aim of this study was to test the hypothesis that VitD3, 25OHD3 and VitD2 affected vitamin D status equally in humans and if rejected, to estimate the difference in activity.

Design: This study was designed as a 3 x 6 weeks (with 4 weeks run-in) double-blinded randomized cross-over study with 12 young, apparently healthy male volunteers and was performed during wintertime at 55 degree N. during the 4 weeks run-in period all volunteers received 10 ug/d VitD3 in order to achieve steady-state in vitamin D status. During the 3x6 weeks intervention periods the subjects received 10 ug/d VitD3, 10 ug/d 25OHD3 or 10 ug/d VitD2 in random order. Content of vitD3, VitD2, 25OHD3 and 25-hydroxyvitamin D2 (25OHD2) in serum were quantified my LC-MS/MS using 0.1 mL serum.

DETAILED DESCRIPTION:
A total of 12 apparently healthy, free living male adults aged 20-30 years were recruited in this 3x6 weeks vitamin D intervention trial. Subjects were recruited among students from the University of Copenhagen through the use of advertisements placed around the University of Copenhagen. Volunteers were excluded if they had BMI > 27 kg/m2, had donated blood within the last three month, has any chronic diseases, used medication regularly, hypercalcemic, had excessive alcohol use, known malabsorption syndromes or used medication known to interfere with vitamin D metabolism. Furthermore, to decrease sun exposure, volunteers who planned to go skiing or travel south during the study was excluded. All subjects were Caucasian, had low habitual fish intake (less than twice a week) and were non-smokers. All subjects were instructed to maintain the same level of physical activity throughout the study and agreed to refrain from donating blood, as well as taking any kind of vitamin, mineral or dietary supplement other than supplements provided in the study. All subjects also agreed to abstain from taking solarium during the intervention. The study was approved by The Local Research Ethics Committee of Copenhagen and Frederiksberg. All participants gave written consent in accordance with the Helsinki declaration.

Design and conduct of study The present study was designed as a double blinded randomised cross over trial in which adult males were assigned to receive tablets containing 10 µg vitD3, 10 µg 25OHD3 and 10 µg vitD2 in random order. Prior to the intervention all subjects received 10 µg vitD3 for 4 weeks in order to achieve steady state in vitamin D status.

The vitamin D tablets (Jette) Compliance was assessed by tablet counting. The study was carried out in Copenhagen, Denmark (latitude 55 degree N). All subjects were recruited in September and run-in periods started in mid-October and the study was finished at the end of March. During the study the subjects were examined at screening, on day 1, 22 and day 42. Blood sample was collected 5 times; before run-in, at baseline, and at end of period, 1, 2 and 3, respectively. Blood samples were drawn after 12 h fasting, in the morning (between 0800 and 0900) by by a trained medical laboratory technician. Subjects were informed not to drink any kind of alcohol and to abstain from hard physical work 24 h before each blood sampling. They were, however, allowed to drink up to ½ L of water. Blood was collected by venipuncture into 10 ml dry tubes for analysis of serum vitamin D, in 5 ml tubes for analysis of serum PTH and in 7 ml Trace element free tubes for analysis of calcium. Blood samples was kept at 20 degree C and centrifuged after 40 min at 3000 g for 15 min. serum was then transferred into plastic tubes and stored at -80 degree C for vitamin d analysis or -20 degree C for Ca and PTH. Anthropometric measures, including height and weight, were taken at baseline. Body weight was measured to nearest 0.1 kg by use of an electronic decimal weight. Subjects were asked to empty their bladder before measuring weight only wearing underwear. The height was measured to nearest cm with the subject standing without shoes, gathering feeds and the head looking forward in horizontal plan.

Habitual intake of calcium and vitamin D was estimated by using a validated food-frequency questionnaire. A health and lifestyle questionnaire, which assessed habitual fish intake, physical activity, general health, smoking status and alcohol consumption, was completed at screening.

Laboratory analysis Serum 25OHD Serum intact parathyroid hormone Serum total calcium

ELIGIBILITY:
Inclusion Criteria:

* No drug use
* BMI< 25 kg/m2
* Do not eat fish more than 2 x weekly
* Not donated blood within 3 months
* No Holiday plans in Winter 2006-2007

Exclusion Criteria:

* Any disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Serum 25OHD | 1 year
  Vitamin D status after intervention with different types of vitamin D

SECONDARY OUTCOMES:
Serum Parathyreoideahormon | 1 year
  Marker for ca status
Serum Ca | 1 year
  Marker for Ca status

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Bügel, Principal Investigator — Department of Nutrition, Exercise and Sports
Locations (1):
- Department of Nutrition, Exercise and Sports, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes